CLINICAL TRIAL: NCT06018714
Title: The Clinical Efficacy of Modified Fruquintinib as Maintenance Treatment for Colorectal Cancer Liver Metastases After NED: Phase II Single-arm Prospective Study
Brief Title: Efficacy of Modified Fruquintinib in Colorectal Cancer Liver Metastases: A Phase II Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, ZHI-ZHONG PAN, Prof., Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-FXY-096-Department of CRC
Record Dates: First submitted 2023-08-09; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Colorectal Cancer Metastatic
Keywords: Colorectal cancer; Fruquintinib
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-arm, phase II study aimed at exploring the clinical efficacy and safety of fruquintinib as maintenance therapy for advanced CRC patients who achieve NED after adjuvant chemotherapy. Patients will receive full supportive care while on this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fruquintinib group (Experimental): Patients will receive Fruquintinib maintenance treatment for six months, or until tumor recurrence, metastasis, or intolerable drug toxicities occur within six months.
  After achieving no evidence of disease (NED), a chest, abdomen, and pelvic CT scan with contrast or a chest CT scan with abdominal and pelvic MRI scan will be performed every 6 months within 2 years. Colonoscopy will be performed annually. CEA, CA19-9, and abdominal and pelvic ultrasound will be performed every 3 months. If abnormalities are found, further imaging studies and colonoscopy will be conducted, and if necessary, a PET/CT scan will be performed.
  Interventions: Drug: Fruquintinib

INTERVENTIONS:
Drug: Fruquintinib — Drug:
  Maintenance treatment regimen:
  Fruquintinib 5 mg, qd, po, with three weeks of continuous treatment followed by one week of drug discontinuation. Each treatment cycle lasts four weeks. The treatment will be continued for six months, or until tumor recurrence, metastasis, or intolerable drug toxicities occur within six months.
  Adverse drug reactions that occur during the trial will be graded according to the NCI CTCAE version 5.0 and dose adjustments will be made according to the corresponding rules.

SUMMARY:
The overall 5-year survival rate for patients with colorectal liver metastases (CRLM) is still less than 20%. Surgery-based local treatment can achieve no evidence of disease (NED) in CRLM patients, but over 60% of patients experience recurrence even after achieving NED. Even with adjuvant therapy for the 6-month perioperative period after achieving NED, the recurrence rate remains high. Fruquintinib is a selective anti-angiogenic inhibitor that may help reduce tumor recurrence and prolong the time to recurrence and metastasis. The Chinese Society of Clinical Oncology (CSCO) guidelines have recommended fruquintinib as a third-line therapy for colorectal cancer. This study aims to evaluate the effectiveness and safety of fruquintinib as a maintenance therapy for patients with advanced colorectal cancer (CRC) who have achieved no evidence of disease (NED) after completing adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. . The pathological diagnosis was colorectal adenocarcinoma liver metastasis；
2. . Age: 18 to 75 years old,allgenders；
3. . Patients who have previously received first-line chemotherapy and have achieved disease control (PR+SD) according to RECIST 1.1;
4. . Patients with liver metastasis of colorectal cancer who have undergone curative local treatment (surgery, ablation, SBRT) and achieved no evidence of disease (NED). Definition of NED: a. After local treatment, no residual signs of primary or metastatic tumors are observed on CT, MRI, PET-CT imaging, or b. No cancer cells are found in biopsies of suspicious lesions；
5. .Completed adjuvant chemotherapy after achieving NED (e.g. 4-8 cycles of CapOX regimen, 6-12 cycles of FOLFOX regimen, or without receiving adjuvant chemotherapy recently) and evaluated as no disease progression. Last chemotherapy within 2 months from enrollment.
6. . The time interval between the last chemotherapy and enrollment does not exceed 2 months;
7. . Performance status (ECOG score) ≤ 2
8. . Hematology: WBC > 3 × 10^9 / L; PLT > 80 × 10^9 / L; Hb > 90 g/L;
9. . Liver function: ALT and AST ≤ 2.5 × ULN; bilirubin ≤ 1.5 × ULN;
10. .Renal function: Serum creatinine ≤ 1.5 × ULN or creatinine clearance rate (CCr) ≥ 60 ml/min;
11. .Signed informed consent, willingness to undergo treatment according to this protocol, and good compliance with medication.

Exclusion Criteria:

1. .Patients with tumor progression before enrollment following the completion of chemotherapy.
2. .Intestinal obstruction or incomplete intestinal obstruction.
3. .Co-existing with other serious illnesses, including severe electrolyte disorders, bleeding tendencies, etc.
4. .Active or uncontrolled severe infections: a) Known human immunodeficiency virus (HIV) infection. b) Known clinically significant liver disease history, including viral hepatitis [known carriers of hepatitis B virus (HBV) must exclude active HBV infection, i.e., HBV DNA positive (>1×104 copies/mL or >2000 IU/mL)]. c) Known hepatitis C virus (HCV) infection with positive HCV RNA (>1×103 copies/mL), or other hepatitis, liver cirrhosis.
5. .Women who are pregnant or breastfeeding and have childbearing potential but are not taking adequate contraceptive measures.
6. .Patients with severe brain disorders or mental illnesses (such as depression, mania, obsessive-compulsive disorder, and schizophrenia) that affect the patient's ability to self-report.
7. .Patients with autoimmune diseases, blood system disorders, and a history of organ transplantation, long-term use of steroids, or immunosuppressive agents.
8. .History of other malignant tumors within the past 5 years, excluding cured cervical carcinoma in situ or basal cell carcinoma of the skin.
9. .History of organ transplantation (including autologous bone marrow transplantation and peripheral stem cell transplantation).
10. .Known or suspected allergies to the investigational drug fruquintinib.
11. .Hypertension that cannot be well controlled with antihypertensive medications (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg).
12. .Active cardiac disease within 6 months prior to treatment, including myocardial infarction, severe/unstable angina pectoris. Left ventricular ejection fraction <50% on echocardiography, poorly controlled arrhythmias.
13. .Urinalysis indicating urine protein ≥2+ and 24-hour urine protein quantification >1.0g.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
2-year recurrence and metastasis rate | 2 years after NED
  To evaluate the clinical efficacy and safety of fruquintinib as maintenance therapy for advanced CRC patients who achieve NED after adjuvant chemotherapy, with the 2-year recurrence and metastasis rate as the primary indicator.

SECONDARY OUTCOMES:
2-year disease-free survival rate | 2 years after NED
  To evaluate 2-year recurrence-free survival rate, 2-year overall survival rate, recurrence-free survival period in patients accepting fruquintinib maintenance therapy.

OTHER OUTCOMES:
completion rate of maintenance therapy | 2 years after NED
  To evaluate safety and completion rate of maintenance therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Colorectal Department,SunYat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No